CLINICAL TRIAL: NCT02984098
Title: 40% Orally Administered Dextrose Gel is More Effective Than 25% Dextrose But Not Sufficiently Reliefs Acute Pain in Term Neonates: A Randomized Controlled Trial
Brief Title: 40% Orally Administered Dextrose Gel is More Effective Than 25% Dextrose
Acronym: 40%D-N-PP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Targu Mures, Romania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POSDRU/159.5/S/133377
Record Dates: First submitted 2016-11-16; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-11

CONDITIONS: Acute Pain
Keywords: procedural pain, 40% Dextrose, heel lance
MeSH Terms: conditions — Acute Pain; Pain, Procedural | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dextrose gel 40% (Experimental): before heel lance, 2 ml oral dextrose gel 40% was administered, and pain related intensity was evaluated with premature infant pain profile scale
  Interventions: Drug: Dextrose
- Dextrose gel 25% (Active Comparator): before heel lance, 2ml oral dextrose gel 25% was administered, and pain related intensity was evaluated with premature infant pain profile scale
  Interventions: Drug: Dextrose

INTERVENTIONS:
Drug: Dextrose — before heel lance, 2ml oral dextrose gel 25%or 40% was administered, and pain related intensity was evaluated with premature infant pain profile scale

SUMMARY:
The aim of this study was to evaluate the safe of 40% Dextrose oral administration on blood glucose concentration and to reducing of pain before painful procedures on healthy term neonate 72 hours aged.

DETAILED DESCRIPTION:
During the study period around 2000 term neonates were born in the university affiliated hospital. Five to 7 term neonates were assessed weekly by the principal investigator (PI) for study eligibility. The parents of neonates who met the inclusion criteria received information about the study after which they were invited to participate. Written informed consent from parent was obtained. The PI entered data into the online Research Randomizer which provided a randomization number corresponding to a numbered treatment pack containing two syringes, each containing 2ml of an identical and therefore blinded liquid. Study investigators, clinical staff, parents and monitors remained blinded to treatment allocation until data analysis was completed. To ensure standardization the included term infants were not breastfeed 30' prior to the heel stick and a standardized heel lance was used.Each infant was taken to a separate room with the mother by the assigned nurse to provide a quite environment. All infants were awake at the time of the procedure. Their clothes were removed and wet diapers were changed. In both groups, the infants were placed in a supine position on a changing table. Dextrose administration and the heel stick were undertaken by an experienced staff neonatal nurse. The heel was warmed with a warm wet towel up 2' minutes before the procedure. The heel was disinfected shortly before the procedure started.

ELIGIBILITY:
Inclusion Criteria:

* were born at ≥ 37 weeks of gestation were
* APGAR score of ≥ 7 five minutes after birth
* had a postnatal age of ≥ 72 hours
* were breastfed (but not 30' prior to the testing HS)
* were undergoing a routine heel stick for metabolic screening between the third and fifth postnatal day

Exclusion Criteria:

* any kind of medical instabilities needing a transfer to the neonatal intensive care unit (NICU)
* severe intrapartum asphyxia defined as a 5' Apgar score less than 3
* parenteral nutrition and the presence of neurological symptoms
* congenital anomalies
* other conditions requiring treatment for hypo- or hyperglycemia
* those in which the heel lance procedure failed

Ages: 3 Days to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pain reactivity changes after orally administered 0.5 ml/ kg body 40% dextrose gel or 25% dextrose as procedural pain relief in term neonates requiring a routine heel stick 72 hours after birth. | one routine heel stick 72 hours after birth
  Pain reactivity changes were assessed using the Premature Infant Pain Profile-revised (PIPP-R scale) which is composed of three behavioral, two physiological and two contextual pain indicators. Five measurements were undertaken during one routine heel stick which took place 72 hours after birth, on the bed side and coded through direct observation during 15 seconds at 5 different time points:
  1. t0: before the heel lance (= baseline 30 minutes without stimuli before heel stick);
  2. t1: at the end of the heel lance (after the ending of the squeezing of the heel and successful collection of blood drops);
  3. t2: at 1 minute recovery time;
  4. t3: at 2 minutes recovery time;
  5. t4: at 5' minutes recovery time.

SECONDARY OUTCOMES:
Blood glucose levels changes after orally administered 0.5 ml/kg body 40% dextrose gel or 25% dextrose as procedural pain relief in term neonates requiring a routine heel stick 72 hours after birth. | one routine heel stick 72 hours after birth and at 30 minutes after orally 0.5 ml/kg body 40% dextrose gel or 25% dextrose
  Blood glucose levels were measured at two different time points:
  1. First glucose level measurement was performed during heel stick by means of the last drop of collected blood
  2. Second glucose level measurement was performed 30 minutes after the heel stick.

CONTACTS AND LOCATIONS:
Overall Officials: LAURA MIHAELA SUCIU, MD,PhD, Principal Investigator — University of Targu Mures, Romania
Locations (1):
- Department of Pediatrics, University of Medicine and Pharmacy Tirgu Mures, Târgu Mureş, Romania

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Carbajal R, Rousset A, Danan C, Coquery S, Nolent P, Ducrocq S, Saizou C, Lapillonne A, Granier M, Durand P, Lenclen R, Coursol A, Hubert P, de Saint Blanquat L, Boelle PY, Annequin D, Cimerman P, Anand KJ, Breart G. Epidemiology and treatment of painful procedures in neonates in intensive care units. JAMA. 2008 Jul 2;300(1):60-70. doi: 10.1001/jama.300.1.60. PMID 18594041
- [Background] Stevens BJ, Abbott LK, Yamada J, Harrison D, Stinson J, Taddio A, Barwick M, Latimer M, Scott SD, Rashotte J, Campbell F, Finley GA; CIHR Team in Children's Pain. Epidemiology and management of painful procedures in children in Canadian hospitals. CMAJ. 2011 Apr 19;183(7):E403-10. doi: 10.1503/cmaj.101341. Epub 2011 Apr 4. PMID 21464171
- [Background] Cignacco E, Hamers JP, van Lingen RA, Zimmermann LJ, Muller R, Gessler P, Nelle M. Pain relief in ventilated preterms during endotracheal suctioning: a randomized controlled trial. Swiss Med Wkly. 2008 Nov 1;138(43-44):635-45. doi: 10.4414/smw.2008.12288. PMID 19005869
- [Background] Roofthooft DW, Simons SH, Anand KJ, Tibboel D, van Dijk M. Eight years later, are we still hurting newborn infants? Neonatology. 2014;105(3):218-26. doi: 10.1159/000357207. Epub 2014 Feb 4. PMID 24503902
- [Background] Anand KJ, Scalzo FM. Can adverse neonatal experiences alter brain development and subsequent behavior? Biol Neonate. 2000 Feb;77(2):69-82. doi: 10.1159/000014197. PMID 10657682
- [Background] Anand KJ. Pain, plasticity, and premature birth: a prescription for permanent suffering? Nat Med. 2000 Sep;6(9):971-3. doi: 10.1038/79658. No abstract available. PMID 10973310
- [Background] Harrison D, Yamada J, Stevens B. Strategies for the prevention and management of neonatal and infant pain. Curr Pain Headache Rep. 2010 Apr;14(2):113-23. doi: 10.1007/s11916-009-0091-0. PMID 20425200
- [Background] Wilkinson DJ, Savulescu J, Slater R. Sugaring the pill: ethics and uncertainties in the use of sucrose for newborn infants. Arch Pediatr Adolesc Med. 2012 Jul 1;166(7):629-33. doi: 10.1001/archpediatrics.2012.352. PMID 22751876
- [Background] Stevens B, Yamada J, Ohlsson A. Sucrose for analgesia in newborn infants undergoing painful procedures. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD001069. doi: 10.1002/14651858.CD001069.pub3. PMID 20091512
- [Background] COMMITTEE ON FETUS AND NEWBORN and SECTION ON ANESTHESIOLOGY AND PAIN MEDICINE. Prevention and Management of Procedural Pain in the Neonate: An Update. Pediatrics. 2016 Feb;137(2):e20154271. doi: 10.1542/peds.2015-4271. Epub 2016 Jan 25. PMID 26810788
- [Background] Harrison D, Beggs S, Stevens B. Sucrose for procedural pain management in infants. Pediatrics. 2012 Nov;130(5):918-25. doi: 10.1542/peds.2011-3848. Epub 2012 Oct 8. PMID 23045554
- [Background] Bueno M, Yamada J, Harrison D, Khan S, Ohlsson A, Adams-Webber T, Beyene J, Stevens B. A systematic review and meta-analyses of nonsucrose sweet solutions for pain relief in neonates. Pain Res Manag. 2013 May-Jun;18(3):153-61. doi: 10.1155/2013/956549. PMID 23748256
- [Background] Harrison D, Bueno M, Yamada J, Adams-Webber T, Stevens B. Analgesic effects of sweet-tasting solutions for infants: current state of equipoise. Pediatrics. 2010 Nov;126(5):894-902. doi: 10.1542/peds.2010-1593. Epub 2010 Oct 11. PMID 20937658
- [Background] Stevens B, Yamada J, Beyene J, Gibbins S, Petryshen P, Stinson J, Narciso J. Consistent management of repeated procedural pain with sucrose in preterm neonates: Is it effective and safe for repeated use over time? Clin J Pain. 2005 Nov-Dec;21(6):543-8. doi: 10.1097/01.ajp.0000149802.46864.e2. PMID 16215340
- [Background] Lefrak L, Burch K, Caravantes R, Knoerlein K, DeNolf N, Duncan J, Hampton F, Johnston C, Lockey D, Martin-Walters C, McLendon D, Porter M, Richardson C, Robinson C, Toczylowski K. Sucrose analgesia: identifying potentially better practices. Pediatrics. 2006 Nov;118 Suppl 2:S197-202. doi: 10.1542/peds.2006-0913R. PMID 17079623
- [Background] Gaspardo CM, Miyase CI, Chimello JT, Martinez FE, Linhares MBM. Is pain relief equally efficacious and free of side effects with repeated doses of oral sucrose in preterm neonates? Pain. 2008 Jul;137(1):16-25. doi: 10.1016/j.pain.2007.07.032. Epub 2007 Sep 12. PMID 17854995
- [Background] Johnston CC, Filion F, Snider L, Limperopoulos C, Majnemer A, Pelausa E, Cake H, Stone S, Sherrard A, Boyer K. How much sucrose is too much sucrose? Pediatrics. 2007 Jan;119(1):226. doi: 10.1542/peds.2006-3001. No abstract available. PMID 17200300
- [Background] Bellieni CV, Stazzoni G, Tei M, Alagna MG, Iacoponi F, Cornacchione S, Bertrando S, Buonocore G. How painful is a heelprick or a venipuncture in a newborn? J Matern Fetal Neonatal Med. 2016;29(2):202-6. doi: 10.3109/14767058.2014.992334. Epub 2014 Dec 23. PMID 25534000
- [Background] Cignacco E, Hamers JP, Stoffel L, van Lingen RA, Schutz N, Muller R, Zimmermann LJ, Nelle M. Routine procedures in NICUs: factors influencing pain assessment and ranking by pain intensity. Swiss Med Wkly. 2008 Aug 23;138(33-34):484-91. doi: 10.4414/smw.2008.12147. PMID 18726734
- [Background] Codipietro L, Ceccarelli M, Ponzone A. Breastfeeding or oral sucrose solution in term neonates receiving heel lance: a randomized, controlled trial. Pediatrics. 2008 Sep;122(3):e716-21. doi: 10.1542/peds.2008-0221. PMID 18762508
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Gibbins S, Stevens BJ, Yamada J, Dionne K, Campbell-Yeo M, Lee G, Caddell K, Johnston C, Taddio A. Validation of the Premature Infant Pain Profile-Revised (PIPP-R). Early Hum Dev. 2014 Apr;90(4):189-93. doi: 10.1016/j.earlhumdev.2014.01.005. Epub 2014 Feb 1. PMID 24491511
- [Background] Ballantyne M, Stevens B, McAllister M, Dionne K, Jack A. Validation of the premature infant pain profile in the clinical setting. Clin J Pain. 1999 Dec;15(4):297-303. doi: 10.1097/00002508-199912000-00006. PMID 10617258